CLINICAL TRIAL: NCT06507553
Title: A Translational Phase I, Randomized, Parallel-group, Multi-arm Study to Evaluate Safety and Immunogenicity of an Influenza Vaccine Formulation Containing an Additional H3 Antigen in Healthy Adult Participants 18 to 49 Years of Age and 60 Years of Age and Older.
Brief Title: Study of Influenza Vaccines Containing an Additional H3 Antigen in Healthy Adult Participants 18 to 49 Years of Age and 60 Years of Age and Older
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FBP00005; U1111-1299-2000 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-07-11; First posted 2024-07-18 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Influenza; Healthy Volunteers
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Modified double-blind (observer-blind; blinded for participants and sites, except for those preparing/administering study intervention, and for the Sponsor, except for dedicated Sponsor staff who will be unblinded for interim analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Group 1 (Stage 1) (Active Comparator): Trivalent-Darwin standard dose (SD) formulation will be administered in a single injection to participants aged 18 to 49 years old
  Interventions: Biological: Trivalent-Darwin influenza vaccine
- Group 2 (Stage 1) (Experimental): Augment-Tasmania SD formulation will be administered in a single injection to participants aged 18 to 49 years old
  Interventions: Biological: Augment-Tasmania influenza vaccine
- Group 3 (Stage 1) (Experimental): TIV-2X Darwin SD formulation will be administered in a single injection to participants aged 18 to 49 years old
  Interventions: Biological: TIV-2X Darwin influenza vaccine
- Group 4 (Stage 1) (Experimental): Trivalent-Tasmania SD formulation will be administered in a single injection to participants aged 18 to 49 years old
  Interventions: Biological: Trivalent-Tasmania influenza vaccine
- Group 5 (Stage 2) (Active Comparator): Trivalent-Darwin high dose (HD) formulation will be administered in a single injection to participants of 60 years and older
  Interventions: Biological: Trivalent-Darwin influenza vaccine
- Group 6 (Stage 2) (Experimental): Augment-Tasmania HD formulation will be administered in a single injection to participants of 60 years and older
  Interventions: Biological: Augment-Tasmania influenza vaccine
- Group 7 (Stage 2) (Experimental): TIV-2X Darwin HD formulation will be administered in a single injection to participants of 60 years and older
  Interventions: Biological: TIV-2X Darwin influenza vaccine
- Group 8 (Stage 2) (Experimental): Trivalent-Tasmania HD formulation will be administered in a single injection to participants of 60 years and older
  Interventions: Biological: Trivalent-Tasmania influenza vaccine

INTERVENTIONS:
Biological: Trivalent-Darwin influenza vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Arms: Group 1 (Stage 1); Group 5 (Stage 2)
Biological: Augment-Tasmania influenza vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Arms: Group 2 (Stage 1); Group 6 (Stage 2)
Biological: TIV-2X Darwin influenza vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Arms: Group 3 (Stage 1); Group 7 (Stage 2)
Biological: Trivalent-Tasmania influenza vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Arms: Group 4 (Stage 1); Group 8 (Stage 2)

SUMMARY:
Study FBP00005 is planned to be a translational Phase I, randomized, modified double-blind, active-controlled, multi-center study to be conducted in 2 stages in approximately 400 adults, 18 to 49 years of age and ≥ 60 years of age, in Australia. The purpose of the study is to evaluate the safety and immunogenicity of an influenza vaccine formulation composed of the WHO-recommended virus strains plus an additional H3 strain, compared to formulations containing a single strain from each influenza virus subtype.

Younger adults 18 to 49 years of age will be enrolled in Stage 1 and offered study vaccine formulations at the standard dose. Adults ≥ 60 years of age in Stage 2 will be offered study vaccine formulations at a higher dose.

Enrollment of participants in Stage 2 will occur after review of, and be guided by, safety and immunogenicity results from Stage 1. The study duration will be approximately 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 49 years (Stage 1) or 60 years of age and older (Stage 2) on the day of inclusion
* Participants who are healthy as determined by medical evaluation including medical history and physical examination, if deemed necessary
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, or surgically sterile OR
  * Is of childbearing potential and agrees to use an effective contraceptive method from at least 4 weeks prior to study intervention administration until at least 3 weeks after study intervention administration
* A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) before the first dose of study intervention.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* History of clinically- or laboratory-confirmed diagnosis of influenza infection in the last 12 months
* Known systemic hypersensitivity to any of the study intervention components, or history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular injection, based on investigator's judgment
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (temperature ≥ 38.0°C) on the day of study intervention administration. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Self-reported or prior documented seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C
* Body mass index of 40 or higher
* Current or past diagnosis, personal or in the family, of Guillain-Barré syndrome
* Have known or recently active (within 12 months) neoplastic disease or a current or past diagnosis of any hematologic malignancy
* Receipt of any vaccine in the 4 weeks preceding the study intervention administration or planned receipt of any vaccine in the 3 weeks (approximately 21 days, or until the end of study participation) following study intervention administration
* Previous vaccination against influenza (in the year 2024) with an investigational or marketed vaccine. In the case of adults ≥ 60 years of age (Stage 2 of the study), previous vaccination within 6 months' time period will apply.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Any change in chronic prescription medication or change in medication dose or dosage in the 60 days prior to enrollment

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with immediate adverse event | Within 30 minutes after vaccination
  Includes unsolicited systemic adverse events (or) medically relevant unsolicited systemic adverse events, including those related to the product administered
Number of participants with solicited injection site reactions | Within 7 days after vaccination
  Adverse reactions prelisted in the participant diary
Number of participants with solicited systemic reactions | Within 7 days after vaccination
  Adverse reactions prelisted in the participant diary
Number of participants with unsolicited adverse events | Throughout the study, approximately 3 weeks
  Adverse events other than solicited reactions
Number of participants with serious adverse events | Throughout the study, approximately 3 weeks
  SAEs occurring throughout the study
Number of participants with adverse events of special interest (AESIs) | Throughout the study, approximately 3 weeks
  AESIs occurring throughout the study

SECONDARY OUTCOMES:
Seroconversion based on hemagglutination inhibition antibody titer | Day 1 and day 22
  Seroconversion (HAI Ab titer < 10 [1/dilution] at day 1 and post-injection titer ≥ 40 [1/dilution] at day 22, or titer ≥ 10 [1/dilution] at day 1 and a ≥ 4-fold increase in titer [1/dilution] at day 22)
Seroprotection based on hemagglutination inhibition antibody titer | Day 1 and day 22
  Seroprotection (HAI Ab titer ≥ 40 [1/dilution])
Obtained hemagglutination inhibition antibody titers | Day 1 and day 22
  Assessment of hemagglutination inhibition (HAI) antibody (Ab) titers obtained on day 1 and day 22 after vaccination
Obtained virus neutralization antibody titers | Day 1 and day 22
  Assessment of virus neutralization (VN) antibody (Ab) titers obtained on day 1 and day 22 after vaccination
Individual hemagglutination inhibition titers ratio | Day 1 and day 22
  Seroconversion (HAI Ab titer < 10 [1/dilution] at day 1 and post-injection titer ≥ 40 [1/dilution] at day 22, or titer ≥ 10 [1/dilution] at day 1 and a ≥ 4-fold increase in titer [1/dilution] at day 22)
Individual virus neutralization titers ratio | Day 1 and day 22
  Individual VN titers ratio (day 22/ day 1)
2-fold rise in virus neutralization titers | From day 1 to day 22
4-fold rise in virus neutralization titers | From day 1 to day 22

CONTACTS AND LOCATIONS:
Locations (10):
- Australia (10):
  - Investigational Site Number : 0360002, Botany, New South Wales
  - Investigational Site Number : 0360010, Brookvale, New South Wales
  - Investigational Site Number : 0360012, Maroubra, New South Wales
  - Investigational Site Number : 0360011, Miranda, New South Wales
  - Investigational Site Number : 0360004, Sippy Downs, Queensland
  - Investigational Site Number : 0360003, Southport, Queensland
  - Investigational Site Number : 0360013, Taringa, Queensland
  - Investigational Site Number : 0360007, Adelaide, South Australia
  - Investigational Site Number : 0360001, Melbourne, Victoria
  - Investigational Site Number : 0360005, Morayfield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: FBP00005 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26051&tenant=MT_SNY_9011